CLINICAL TRIAL: NCT03773562
Title: Imaging the Migraine Brain Pre- and Post-Erenumab: an MRI Study to Identify Functional and Structural Changes That Correlate With Patient Improvement
Brief Title: Imaging the Migraine Brain Pre- and Post-Erenumab
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001497
Record Dates: First submitted 2018-11-27; First posted 2018-12-12 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Migraine
Keywords: Migraine; Magnetic Resonance Imaging; Brain Structure; Brain Function
MeSH Terms: conditions — Migraine Disorders | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Erenumab (Other): All participants receive erenumab 140mg by subcutaneous injection at baseline and again 4 weeks later.
  Interventions: Drug: Erenumab

INTERVENTIONS:
Drug: Erenumab — Erenumab will be used per label instructions.
  Other Names: Aimovig

SUMMARY:
Researchers are trying to determine if there is a difference between brain images of subjects that do respond to treatment with erenumab and subjects who do not respond to treatment with erenumab using Magnetic Resonance Imaging (MRI).

ELIGIBILITY:
Inclusion Criteria

* 18-65 years of age
* Episodic migraine (with or without aura) or chronic migraine according to the diagnostic criteria included within the International Classification of Headache Disorders 3 (ICHD-3)
* 6-25 migraine days per month on average over the 3 months prior to screening, confirmed by run-in phase prospective data collection
* Duration since migraine onset of at least 12 months prior to screening based on medical records and/or patient self-report

Exclusion Criteria

* Older than 50 years of age at migraine onset
* History of cluster headache or hemiplegic migraine
* Continuous headache pain (i.e. no pain-free periods of any duration during the one month before screening)
* Opioid- or butalbital-containing analgesics on 6 or more days per month during the 2 months prior to the start of the baseline phase
* History of major psychiatric disorder such as schizophrenia and bipolar disorder
* History or evidence of any unstable or clinically significant medical condition, that in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* No therapeutic response in migraine prevention after an adequate therapeutic trial of 4 or more of the following medication categories: Category 1- divalproex sodium, sodium valproate; Category 2- topiramate; Category 3- beta-blockers; Category 4- tricyclic antidepressants; Category 5- venlafaxine or desvenlafaxine, duloxetine or milnacipran; Category 6- flunarizine, verapamil; Category 7- lisinopril, candesartan; Category 8- botulinum toxin. No therapeutic response is defined as no reduction in headache frequency, duration, or severity after administration of the medication for at least 6 weeks at the generally accepted therapeutic dose(s) based on the investigator's assessment. Lack of sustained response to a medication and failure to tolerate a therapeutic dose are not considered to be "no therapeutic response".
* Concomitant use of 3 or more of the following medications for migraine prevention within 2 months before the start of the baseline phase or throughout the study: divalproex sodium, sodium valproate, topiramate, carbamazepine, gabapentin, beta-blockers, tricyclic antidepressants, venlafaxine, desvenlafaxine, duloxetine, milnacipran, flunarizine, verapamil, lomerizine, lisinopril, candesartan, clonidine, guanfacine, cyproheptadine, methysergide, pizotifen, butterbur, feverfew, magnesium (at least 600 mg per day), riboflavin (at least 100 mg per day). Use of up to two medications is permitted as long as the dose has been stable for at least 2 months before the start of the run-in phase and during the study.
* Botulinum toxin (in the head and/or neck region) within 4 months before the start of the baseline phase and throughout the study
* Ergotamine derivatives, steroids, and triptans used for migraine prophylaxis within 2 months before the start of the baseline phase and throughout the study
* Procedures (e.g. nerve blocks) used for migraine prophylaxis within 2 months before the start of the baseline phase and throughout the study
* History of myocardial infarction, stroke, transient ischemic attack, unstable angina, coronary artery bypass surgery, or other revascularization procedures within 12 months prior to screening.
* Contraindications to MRI including, but not limited to: Metal implants, aneurysm clips, severe claustrophobia, implanted electronic devices, insulin or infusion pump, cochlear/otologic/ear implant, non-removable prosthesis, implanted shunts/catheters, certain intrauterine devices, tattooed makeup, body piercings that cannot be removed, metal fragments, wire sutures or metal staples.
* Factors that Reduce MR Image Quality and Interpretability: dental braces or other non-removable devices (e.g. retainers); prior brain surgery; known brain MRI abnormality that in the investigator's opinion will significantly impact MRI data
* Sensory disorders that in the investigator's opinion might affect perception of cutaneous thermal stimuli (e.g. peripheral neuropathy)
* Pregnancy
* Lactation
* Not willing to use a reliable form of contraception (for women of childbearing potential) through 16 weeks after the last dose of erenumab. Acceptable methods of birth control include not having intercourse, hormonal birth control methods, intrauterine devices, surgical contraceptive methods, or two barrier methods (each partner must use a barrier method) with spermicide. A reliable form of contraception must be started prior to or at the time of starting the run-in phase. Not being of childbearing potential is defined as any woman who: 1) is post-menopausal by history, defined as: a) At least 55 years of age with cessation of menses for 12 or more months, OR b) Younger than 55 years of age but no spontaneous menses for at least 2 years, OR c)Younger than 55 years of age and spontaneous menses within the past 1 year, but currently amenorrheic (e.g. spontaneous or secondary to hysterectomy), AND with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels at least 40 IU/L) or postmenopausal estradiol level (less than 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved, OR d) Underwent bilateral oophorectomy, OR e) Underwent hysterectomy, OR f) Underwent bilateral salpingectomy
* Currently receiving treatment in another drug study or an investigational device study, or less than 90 days prior to screening since ending treatment on another investigational device or drug study(-ies)
* Has received calcitonin gene-related peptide (CGRP) monoclonal antibody within 4 months of the start of the run-in phase
* Active chronic pain condition that in the investigator's opinion is unrelated to migraine (e.g. chronic pelvic pain)
* Acute pain condition that in the investigator's opinion is unrelated to migraine (e.g. post-surgical pain)
* Unable to provide informed consent
* Less than 80% compliance with providing headache diary data during the run-in phase (i.e. provides data on less than 80% of days)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd J Schwedt, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schwedt TJ, Nikolova S, Dumkrieger G, Li J, Wu T, Chong CD. Longitudinal changes in functional connectivity and pain-induced brain activations in patients with migraine: a functional MRI study pre- and post- treatment with Erenumab. J Headache Pain. 2022 Dec 14;23(1):159. doi: 10.1186/s10194-022-01526-5. PMID 36517767
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erenumab
Started | 50
Completed | 29
Not Completed | 21
Not completed — Did not have 6-25 migraine days during run-in | 10
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erenumab
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 41
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Resting State Functional Connectivity
Description: Brain MRI resting state functional connectivity measured as global efficiency percentage. An increase in global efficiency suggests an improvement in the ability of the brain regions to functionally communicate on a global scale. Efficiency relates to the network. In this case, the investigators defined the network to be the pain matrix. Increased efficiency would mean the connectivity within the matrix is increased and more efficient. This has not been attributed to a clinical outcome but is rather a characteristic of the network.
Time Frame: 8 weeks
Population: Of the 32 participants to complete a functional MRI (fMRI) of the brain, 18 participants were identified as erenumab responders and 14 were erenumab non-responders.
Measure: Mean (Standard Error); unit: global efficiency percentage
Arm/Group | Erenumab
Number analyzed (Participants) | 32
global efficiency percentage
  Erenamab responders: number analyzed (Participants) | 18
  Erenamab responders | 26.2 (1.1)
  Erenumab non-responders: number analyzed (Participants) | 14
  Erenumab non-responders | 23.3 (0.7)
Statistical Analysis 1: Comparison: Erenumab; Responders vs Non-responders; Test type: Superiority; p = 0.04, t-test, 2 sided

2. Secondary Outcome: Erenumab Responders
Description: The number of participants who responded to erenumab treatment. Treatment response was defined as at least a 50% reduction in the frequency of migraine days during weeks 5-8 compared to the 4 week pre-treatment run-in phases as recorded in the headache diary.
Time Frame: 8 weeks
Population: Of the 50 participants enrolled, 32 received erenumab treatment and completed a functional MRI (fMRI) of the brain.
Measure: Count of Participants; unit: Participants
Arm/Group | Erenumab
Number analyzed (Participants) | 32
Participants | 18

3. Secondary Outcome: Iron Accumulation in Periaqueductal Gray Brain Region
Description: Iron accumulation in the periaqueductal gray as measured by magnetic resonance imaging (MRI) transverse relaxation rates (T2*).
Time Frame: 8 weeks
Population: Of the 28 participants with complete MRI T2* results, 15 participants were identified as erenumab responders and 13 were erenumab non-responders.
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | Erenumab
Number analyzed (Participants) | 28
milliseconds (ms)
  Erenumab responders: number analyzed (Participants) | 15
  Erenumab responders | 43.0 (1)
  Erenumab non-responders: number analyzed (Participants) | 13
  Erenumab non-responders | 32.5 (1)
Statistical Analysis 1: Comparison: Erenumab; Responders vs Non-Responders; Test type: Superiority; p = 0.002, t-test, 2 sided

4. Secondary Outcome: Iron Accumulation in Anterior Cingulate Cortex Brain Region
Description: Iron accumulation in the anterior cingulate cortex as measured by magnetic resonance imaging (MRI) transverse relaxation rates (T2*).
Time Frame: 8 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: milliseconds (ms)
Arm/Group | Erenumab
Number analyzed (Participants) | 28
milliseconds (ms)
  Erenumab responders: number analyzed (Participants) | 15
  Erenumab responders | 50 (1)
  Erenumab non-responders: number analyzed (Participants) | 13
  Erenumab non-responders | 40 (1)
Statistical Analysis 1: Comparison: Erenumab; Responders vs Non-responders; Test type: Superiority; p = 0.01, t-test, 2 sided

5. Secondary Outcome: Change in the Migraine Disability Assessment Questionnaire (MIDAS)
Description: The MIDAS questionnaire consists of 5 questions that assess the degree of headache related disability. Each question asks the patient to record the number of days in the past 3 months where a headache has impacted various daily life activities. The individual responses to each of the five questions are then added to obtain a total score and level of disability. A total score of 0-5 days reflects little or no disability (Grade I); 6-10 days is mild disability (Grade II); 11-20 days is moderate disability (Grade III) and over 21 days is severe disability (Grade IV). A lower score indicates less disability while a higher score reflects more disability.
Time Frame: Baseline, 8 weeks
Population: Of the 28 participants that completed the MIDAS questionnaire, 15 participants were identified as erenumab responders and 13 were erenumab non-responders.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Erenumab
Number analyzed (Participants) | 28
score on a scale
  Erenumab responders: number analyzed (Participants) | 15
  Erenumab responders | -16.5 (16)
  Erenumab non-responders: number analyzed (Participants) | 13
  Erenumab non-responders | 5.8 (13)

6. Secondary Outcome: ROI-ROI Functional Connectivity of Middle Temporal Left With Supramarginal Gyrus Right Regions of the Brain
Description: Temporal correlations in blood oxygen level dependent (BOLD) signal fluctuations between selected regions of interest (ROIs). The correlation coefficient ( r ) is measured between seed regions. This measurement is bound by the range [ -1 to 1]. In order to perform statistical tests (such as T-tests) we Fisher transform the correlation coefficient from [-1 1] to a real number [ -infinity infinity] Mathematically it is: z=atanh( r ). The Z-score themselves are functional connectivity between the regions and do not serve as clinical biomarkers. The difference, and longitudinal changes are of greater interest as they indicate alterations to normal pain processing. A more efficient pain processing network would suggest that more of these regions are being enlisted and with greater connectivity.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responder: number analyzed (Participants) | 18
  Erenumab responder | 0.34
  Erenumab non-responder: number analyzed (Participants) | 14
  Erenumab non-responder | 0.02
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0003, t-test, 2 sided

7. Secondary Outcome: ROI-ROI Functional Connectivity of Temporal Pole Right With Middle Occipital Right
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responders: number analyzed (Participants) | 18
  Erenumab responders | 0.24
  Erenumab non-responders: number analyzed (Participants) | 14
  Erenumab non-responders | -0.08
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0003, t-test, 2 sided

8. Secondary Outcome: ROI-ROI Functional Connectivity of Inferior Lateral Parietal Right With Middle Frontal Left
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responders: number analyzed (Participants) | 18
  Erenumab responders | -0.07
  Erenumab non-responders: number analyzed (Participants) | 14
  Erenumab non-responders | 0.24
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0003, t-test, 2 sided

9. Secondary Outcome: ROI-ROI Functional Connectivity of Dorsolateral Prefrontal Cortex Left With Hypothalamus Right
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responder: number analyzed (Participants) | 18
  Erenumab responder | 0.02
  Erenumab non-responder: number analyzed (Participants) | 14
  Erenumab non-responder | -0.18
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0033, t-test, 2 sided

10. Secondary Outcome: ROI-ROI Functional Connectivity of Inferior Lateral Parietal Right With Supramarginal Gyrus Right
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responders: number analyzed (Participants) | 18
  Erenumab responders | 0.68
  Erenumab non-responders: number analyzed (Participants) | 14
  Erenumab non-responders | 0.38
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0041, t-test, 2 sided

11. Secondary Outcome: ROI-ROI Functional Connectivity of Ventromedial Prefrontal Cortex Left With Pulvinar Right
Description: as for outcome 6
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: correlation coefficient
Arm/Group | Erenumab
Number analyzed (Participants) | 32
correlation coefficient
  Erenumab responder: number analyzed (Participants) | 18
  Erenumab responder | 0.18
  Erenumab non-responder: number analyzed (Participants) | 14
  Erenumab non-responder | -0.07
Statistical Analysis 1: Comparison: Erenumab; Responder vs non-responder; Test type: Superiority; p = 0.0046, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each participant from the time of the first erenumab treatment through the end of the safety follow up visit (8 weeks after the last dose of the investigational product) for a total of approximately 12 weeks.
Description: Out of 50 participants, 36 received the first dose of erenumab but 4 withdrew from the study prior to completing a function MRI (fMRI) of the brain.
Arm/Group | Erenumab
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 25/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erenumab (N=36)
Dizziness (General disorders) | 3 (3)
Flank pain (General disorders) | 1 (1)
Loss of balance (General disorders) | 1 (1)
Weight gain (General disorders) | 1 (1)
Arm twitching (General disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Agitation (General disorders) | 1 (1)
Communication issues (General disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Covid-19 infection (Infections and infestations) | 1 (1)
Allergic reaction (General disorders) | 1 (1)
West Nile Virus (General disorders) | 1 (1)
Itching/skin sensitivity (General disorders) | 3 (3)
Tinnitus (General disorders) | 1 (1)
Worsening headache (General disorders) | 1 (1)
Constipation (General disorders) | 14 (14)
Abdominal pain (General disorders) | 1 (1)
Injection site erythema (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03773562/Prot_SAP_000.pdf